CLINICAL TRIAL: NCT03835611
Title: Evaluating the Use of a Cognitive Game-Based Treadmill Exercise Program to Improve Balance and Gait in People With Parkinson Disease: A Feasibility Randomized Controlled Trial
Brief Title: Evaluating Effect of Cognitive Game Based Treadmill Exercise Program in Parkinson Disease
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of Recruitment
Sponsor: University of Manitoba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H2018:338
Record Dates: First submitted 2019-01-18; First posted 2019-02-08 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2019-01

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease,; Balance; Gait; Dual Task walking; Feasibility
MeSH Terms: conditions — Parkinson Disease | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Intervention Group: Participants in the intervention group will receive DT TT with GTP. GTP consists of standard treadmill nested with a pressure mapping system and an interactive computer game based sub-station in front of the treadmill. A miniature motion mouse with inbuilt sensors that enables "real-time" movements to be translated in computer sub-station by standard USB will be used. This miniature mouse will be secured to a helmet that participants will wear while walking on the treadmill to interact with computer sub-station. Participants will be expected to play commercial computer games while standing on compliant surface or walking on the treadmill. The motion mouse will help participants to control computer games hand free.
  Interventions: Other: Game based treadmill Platform
- Control Group (Active Comparator): Control group: Participants in the control group will undergo a mixture of current gait training programs available for people with Parkinson Disease. The protocol will be:
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Game based treadmill Platform — The protocol for the intervention group will be:
  * Warm up exercised consisting of rhythmical large movements (10minutes)
  * Dynamic standing balance training by playing commercial games with head rotations while standing on a compliant surface to increase balance demands. (10 Minutes)
  * DT treadmill training, consisting of playing commercial computer games while walking on the treadmill at a self-selected comfortable speed. Participants will be allowed to take rest when required and total effective DT treadmill walking will be for 30minutes. Treadmill speed will be aimed to progress depending on participant performance and documented. An overhead safety harness will always be provided to participants while walking on the treadmill. (25minutes)
  Arms: Intervention group
Other: Control Group — * Warm-up exercise consisting of rhythmical large movements (10 minutes).
  * Core standing balance exercises on a sponge surface (10 minutes).
  * Treadmill walking for 20 minutes, which includes rests periods... An overhead safety harness will be provided to participants while walking on the treadmill
  * Overground walking in an obstacle course. Participants will be instructed to walk along a curved path (marked by tape) and avoid obstacles placed randomly. The obstacle will be thin sponge pads with 10-12 inches in diameter (15minutes).
  Arms: Control Group

SUMMARY:
An inexpensive dual-task gait training protocol has been developed for people with PD namely game based treadmill platform. A feasibility randomized trial clinical trail will be conducted to evaluate the feasibility, acceptability and estimate treatment effect size of the treatment protocol to conduct a future RCT.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is the second most commonly occurring neurological disorder in Canada, affecting approximately 99,000 individuals, and the number is expected to grow to 140,000 individuals by the year 2025. The hallmark of PD pathology is a progressive degeneration of dopaminergic neurons in the basal ganglia (BG). Therefore, there is a significant deterioration of balance and gait function, and especially when concurrently performing a cognitive task (dual-task walking). Fifty percent of individuals with PD also show deficiencies in one or more cognitive area. In addition, up to 80% of PD patients eventually develop dementia. Over 60% of PD, individuals fall each year and a significant portion of those who fall will experience multiple falls. Most falls occur during walking, and the consequences of these falls are often severe, leading to disability, loss of independence (i.e. safe community ambulation). For individuals with PD, community ambulation is strongly associated with the preservation of skills for independent living, leisure/recreational activities, social participation and healthy aging. Daily activities afford numerous situations in which walking must be combined with a cognitive task, such as, navigation, negotiating terrains and obstacles, tracking visual targets, reading, and recall. Walking and cognitive abilities are closely linked, and several studies have demonstrated that walking while performing various cognitive tasks (dual-task walking) results in greater gait disturbances, threats to stability and provokes freezing of gait in PD.

Numerous studies have shown that modest levels of physical activity and targeted physical therapy improves muscle strength, balance, mobility and reduces the risk of falls among older adults. Several studies have also shown improved cognitive function with physical activity, and others report that interventions that enhance cognitive skills led to improvements in fall risk. Because physical and executive cognitive decline both contribute to mobility limitations and an increased fall risk with age, several PD researchers and clinicians have developed balance-walking programs augmented with interactive cognitive activities (Dual-task training). Maximizing participation is also seen as a main goal of interventions. Long-term exercise/training programs are often fraught with low compliance and adherence. An emerging methodology is to combine exercise and activities with computer games, making the training experience more engaging and enjoyable. This approach can be an important tool for rehabilitation because it has the potential to increase participation and exercise adherence. Importantly digital media in the form of computer games can also challenge and train many different aspects of executive cognitive function. For example, many computer games are now readily available in which processing speed, cognitive inhibition, task switching, working memory and problem solving are the main components of the interactive game events.

Based on this information, investigators have has developed and validated an engaging, game-based treadmill platform (GTP), which provides an integrated approach to treat and assess the decline in balance, mobility, Visuomotor and visuospatial executive cognitive function. The GTP consists of 1) a standard treadmill instrumented with a pressure mapping system which to compute several spatiotemporal gait variables and gait stability measures; 2) an innovative interactive computer game subsystem for dual-tasking; and 3) an automated monitoring application which uses advanced data logging and analysis method to record the client's actions and choices while walking and playing targeted cognitive games. Therefore, physical and cognitive performance during exercise can be monitored synchronously and quantified electronically. Proof of principle has been established for the use of the GTP in assessment and treatment of older adult's age70-80 with fall history.

Purpose of this exploratory study is to assess the potential for successful implementation of the novel intervention, predict the feasibility and acceptability of the dual-task exercise program and identify unpredicted harm.

ELIGIBILITY:
Inclusion Criteria:

* Age range 55-70
* Diagnosed with PD according to UK brain bank criteria,
* PD stage 1-3 on Hoehn and Yahr scale,
* On stable medications for PD from past 3months,
* Able to walk 50m independently,
* Montreal Cognitive Assessment( MoCA) score of more than 21(Non-Dementia PD).

Exclusion Criteria:

* Any other neurodegenerative condition,
* Any orthopedic or cardiovascular impairment limiting independent walking for a minimum of 10 minutes.

Ages: 55 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Retention to GTP | 1 year
  Percentage of participants adhering to 10 Weeks of GTP protocol.

SECONDARY OUTCOMES:
Sample size calculation | 1 Year
  Power calculation will be done with coefficient of variation of step length during DT walking as primary outcome measure.

CONTACTS AND LOCATIONS:
Locations (1):
- College of Rehabilitation Sciences, University of Manitoba, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: Undecided
No discussion yet.